### **Protocol**

Study Title: Effect of exercise on the human skeletal muscle

phosphoproteome

**Principal Investigator:** 

Dr. Stuart Phillips<sup>1</sup>

Physician overseeing medical responsibility:

Dr. Steven Baker<sup>3</sup>

**Co-Investigators:** 

Mr Jonathan Mcleod<sup>1</sup>

Mr Aaron Thomas<sup>1</sup>

Dr. Chris McGlory<sup>1</sup>

Dr. Troy Hornberger<sup>2</sup>

# Institution:

<sup>&</sup>lt;sup>1</sup>Department of Kinesiology, McMaster University, Hamilton, Ontario, L8S 4K1, Canada.

<sup>&</sup>lt;sup>2</sup> Department of Comparative Bioscience, University of Wisconsin-Madison, Madison, Wisconsin, 53706, USA

<sup>&</sup>lt;sup>3</sup> Department of Medicine, McMaster University, Hamilton, Ontario, L8S 4K1, Canada.

#### Rationale

Skeletal muscle is a highly plastic tissue, capable of adapting to changes in nutritional intake and contractile activity. For instance, resistance exercise results in a mild stimulation of rates of muscle protein breakdown (MPB) but a greater stimulation of the rates of muscle protein synthesis (MPS) (1-3). When resistance exercise is performed prior to protein ingestion there is a synergistic combination of the two stimuli such that rates of MPS are stimulated over and above those of MPB (4-6). Thus, repeated bouts of resistance exercise, when coupled with protein ingestion, result in the accretion of skeletal muscle protein referred to as hypertrophy (7). Importantly, by changing the nature of the exercise stimulus, it is possible to redirect the focus of the type of skeletal muscle proteins that are being synthesised. For example, we know that prolonged and repeated lower-load dynamic stimulation of skeletal muscle (i.e., endurance exercise training) results in an increase in the expression of mitochondrial genes (8), proteins (8-10), and ultimately enhanced mitochondrial content (11), leading to a shift towards an oxidative phenotype, and improved fatigue resistance (12). Resistance exercise training also stimulates the transcription of genes and accrual of new muscle proteins (13, 14), but these genes and proteins are largely associated with the myofibrillar protein fraction, and regular resistance exercise leads to muscle hypertrophy and increased force-generating capacity (15, 16). However, during the early stages of exercise training, particularly in training-naïve participants there is a significant increase in the expression of genes common to both modalities of exercise (17, 18). It is only with sustained exercise training that there is a 'fine tuning' of the transcriptome, the protein synthetic response, and then the proteome that gives rise to divergent hypertrophic and oxidative phenotypes (17, 19).

# Transcriptional responses to exercise training

Increases in mRNA expression following each exercise session result in enhanced translation of proteins, and ultimately adaptive changes in muscle protein content (12, 19). The temporal pattern of these changes with respect to endurance and resistance exercise training is now becoming clearer. Exerciseinduced mitochondrial biogenesis, for example, is a characteristic feature of endurance exercise training (9, 12, 20) and is underpinned by the coordinated up-regulation of both mitochondrial and nuclear transcripts that encode for proteins involved in the electron transport chain (21-23), and lipid metabolism (24). These transcripts include peroxisome proliferator-activated receptor gamma co-activator (PGC)-1α, nuclear respiratory factors (NRFs), and the mitochondrial transcription factor A (TFAM)(25-27). An acute bout of endurance exercise activates sensors of cellular stress (8, 28), decreases methylation of promoter regions (29), stimulates phosphorylation of mediators of translation initiation (16), and increases the expression of the aforementioned transcripts (PGC-1α, NRFs, TFAM) (8, 12). The transient increase in the expression of genes in the hours following an acute endurance exercise session provides the gene template that precedes the respective increases in protein content observed during exercise training (8, 9). Compared to our understanding of transcriptional responses to endurance training, the corresponding picture with

respect to resistance exercise is relatively less complete. Resistance exercise results in the phosphorylation (i.e., activation) of the mechanistic target of rapamycin complex 1 (mTORC1)(30-33). mTORC1 activation serves to enhance MPS by (1) activating downstream protein kinases such as the ribosomal protein of 70 kDa S6 kinase 1 (p70S6K1) and 4E-binding protein-1 (4EBP1), which subsequently promote ribosomal binding to mRNA to initiate protein synthesis (34-37) and (2) up-regulating the transcription of the translational machinery itself (mRNA, ribosomal content) (38). Thus, resistance exercise stimulates an increase in mTORC1 activity and promotes increases in the rates of myofibrillar MPS through both increased translational efficiency (protein synthesized per unit of mRNA) and translational capacity (the abundance of the translational machinery; ribosomes) (31, 33).

# Posttranslational modification of proteins

Key to exercise-induced adaptation is post-translational modification of proteins. One important post-translational modification is known as phosphorylation. Phosphorylation is the addition of a phosphate group to a target protein by a protein kinase using ATP and Mg (39). The addition of this phosphate can promote the catalytic activity or binding status of a protein resulting in a biological downstream effect. There are over 500 kinases in the human 'kinome'. We (39, 40) and others (16) often assess the phosphorylation status of single or multiple (~ten) kinases/proteins in response to exercise to gain a mechanistic understanding of how exercise alters the skeletal muscle phenotype. However, current methods are largely semi-quantitative (Western blotting) and are biased in terms of which proteins are studied (i.e., the experimenter can only select a limited number of kinases/proteins to measure). Our understanding of how skeletal muscle adaptation is influenced by phosphorylation is therefore limited. Recent developments in mass spectrometry (41, 42) have enabled a wider interrogation of the phosphorylation status of proteins in response to exercise. Indeed, one study, using advanced liquid chromatography-mass spectrometry, revealed 1,004 unique exerciseregulated phosphorylation sites on 562 proteins in human skeletal muscle biopsy samples obtained before and after a bout of endurance exercise (41). This seminal finding has significantly advanced our knowledge regarding how endurance exercise impacts phosphorylation. Yet, no measurements of endpoint MPS were made. Moreover, comparable work has not been performed with resistance exercise. The aim of our investigation is to conduct a similar global phosphoproteomic analysis of skeletal muscle using advanced mass spectrometry following both endurance and resistance exercise in humans. We will also directly measure rates of MPS for the 3 hours following exercise.

The aim of our investigation is to conduct a similar global phosphoproteomic analysis of skeletal muscle using advanced mass spectrometry following resistance and aerobic exercise in humans.

# **Specific Objectives**

- 1. Our primary objective is to examine the effect of resistance exercise on the human skeletal muscle phosphoproteome.
- 2. Our secondary objective is to assess changes in rates of myofibrillar and mitochondrial MPS following resistance and endurance exercise.

# **Hypotheses**

We hypothesize that:

- 1. Both resistance exercise and endurance exercise will result in the widespread phosphorylation of proteins involved in the regulation of energy metabolism, transcription, translation and muscle protein synthesis.
- 2. Resistance exercise will increase myofibrillar MPS to a greater extent than endurance exercise.
- 3. Endurance exercise will increase rates of mitochondrial MPS to a greater extent than resistance exercise.

## **Participants**

#### Inclusion Criteria

In order to participate in this study, participants must be male between the ages of 18 and 30 years <u>and</u> have performed resistance exercise 3 times per week for at least 1 year.

### **Exclusion Criteria**

Participants cannot participate in, or will be released from, this study if they meet <u>one of more</u> of the following criteria:

- Smoker or user of tobacco products
- High physical activity.
- Have health problems such as: renal or gastrointestinal disorders, metabolic disease, heart disease, vascular disease, rheumatoid arthritis, diabetes, poor lung function, uncontrolled blood pressure, dizziness, thyroid problems, or any other health conditions for which you are being treated that might put you at risk for this study.
- Taking anti-diabetic, anti-inflammatory, platelet inhibitor, or anti-coagulant medications.
- Use of an investigational drug product within the last 30 days.
- Have participated in an infusion protocol in the last year.
- Do not understand English or have a condition the PI believes would interfere with a participants' ability to provide informed consent, comply with

the study protocol, or which might confound the interpretation of the study results or put someone at undue risk.

#### Recruitment

Twelve participants (6 male: 6 female) participants will be recruited for this study through poster advertisements. Potential participants will be asked if they meet all of the inclusion criteria and none of the exclusion criteria. During an initial screening visit those who qualify and are interested in participating will be invited to the Exercise Metabolism Research Group (EMRG) laboratory, Ivor Wynne Centre (IWC) at McMaster University to begin testing for the study. The potential participants will then be required to read the Information and Consent Form. A written copy of the consent form will be provided for the participants to read by themselves. Written informed consent will then be obtained.

# Sample Size

This study is an observational pilot investigation. Previous work has detected changes in our primary outcome (phosphoproteome) following endurance exercise with only 4 male participants (41). For the current study, we wish to recruit both male and female participants. Therefore - accounting for participant attrition - we will aim to recruit 12 participants.

# Methodology

A schematic illustration of the experimental design and experimental trial can be seen in Figures 1 and 2, respectively. In a within-subject repeated measures cross-over design, 12 participants (6 male and 6 female) will attend the laboratories at the Dept. of Kinesiology on 6 separate occasions. On the first occasions participants will be assessed for body composition using dual-energy x-ray absorptiometry (DXA) after an overnight fast (~10 hours) followed by familiarization on resistance exercise and endurance exercise equipment. At this point, your two legs will be randomly assigned to the resistance exercise or endurance exercise group.

On the second visit, participants will perform a 1-repetition maximum test on a leg press and leg extension machine. These tests will be used to determine the workload performed on the experimental trials. On the third visit participants will perform a  $V0_{2\,\text{max}}$  test on a cycle ergometer to determine their aerobic fitness. On the same day, subjects will be familiarized with single-leg cycling. On visit 4, subjects will perform another  $V0_{2\text{max}}$  test on a cycle ergometer using one leg only. This test will determine the intensity of cycling performed on the experimental trial. To ensure the intensity is appropriate, the subjects will be familiarized with the experimental trial training programs (see "Exercise protocols" below).

Subjects will then embark on a 3-day period of controlled diet and exercise followed by experimental trials (visits 5 and 6) separated by 1 week. The reason for the two independent trails is that the measurement of MPS requires the

infusion of a stable amino acid isotope (L-[ring-<sup>13</sup>C<sub>6</sub>] phenylalanine), which interferes with the assessment of the phosphoproteome due to the fact they both detect changes in protein mass. Thus the first trial will be conducted to assess exercise-induced changes in the phosphoproteome and the second for MPS, using the L-[ring-<sup>13</sup>C<sub>6</sub>] phenylalanine isotope.

# Acute protocols (Visits 5 + 6)

On visit 5 participants will arrive at the laboratory at approximately 0640 after a 10h overnight fast. After a brief assessment, subjects will rest on a bed for 3 hours. After this period, a skeletal muscle biopsy will be obtained and participants will perform a bout of resistance exercise with a randomised leg, followed by a bout of endurance exercise. Skeletal muscle biopsies will again be obtained immediately following both bouts of exercise and again 3h following exercise. On visit 6, participants will again arrive at the laboratory at approximately 0640 after an overnight fast. This time, a catheter will be placed in the upper forearm. After the placement of the catheter, a primed constant infusion of L-[ring-13C<sub>6</sub>] phenylalanine will be commenced to measure rates of MPS and a catheter placed in the contralateral arm for repeated blood sampling. Exercise and skeletal muscle biopsies will be obtained as in visit 5 (see Figure 2). We have routinely obtained ethical approval and published papers for studies that employ skeletal muscle biopsies and stable amino acid tracers in human volunteers (3, 14, 44-49). Dr. Steven Baker, a liscenced physician, has approved our standard operating procedure and will oversee all muscle biopsy and catheter infusions.



Figure 1 Schematic illustration of experimental design.

R.Ex- 3 sets × 10 reps 70% 1RM leg press followed by leg ext. 2 min recovery between sets and exercises.

E.Ex- 4 × 5 min @ 65% single leg peak power w/ 2.5 min recovery @ 20% peak power.



March 5th 2020

Figure 2. Schematic illustration of Visit 6.

<sup>\*</sup> Timing will change depending on exercise order

#### **Measurements and Measurement Instruments**

# 1 repetition maximum:

The same investigators will administer all strength testing. In short, after a brief general warm-up, a specific warm-up of the given exercise will be performed at approximately 50% of the participant's estimated 1RM based on the 10RM testing. Load will be progressively increased by approximately 10-20% for each repetition until a true 1RM will be reached as previously described (39). Three to 5 min of rest was given between each attempt. A successful attempt required the participant to move the load throughout the full range of motion with correct form.

## VO<sub>2</sub>peak

Subjects will complete double-leg and single-leg incremental peak oxygen uptake (VO<sub>2</sub>peak) tests on a cycle ergometer (Velotron, RacerMate; Seattle, WA). A metabolic cart with an on-line gas collection system (Moxus modular oxygen uptake system, AEI Technologies, Pittsburgh, PA) will acquire oxygen consumption (VO<sub>2</sub>) and carbon dioxide production (VCO<sub>2</sub>) data and heart rate will be monitored continuously with a heart rate monitor (Polar A3, Lake Success, NY). The test will begin with a 1-min warm up at 50 watts (W), after which the power will be increased by 1 W every two seconds until volitional exhaustion or the point at which pedal cadence falls below 60 rpm. Heart rate will be monitored continuously throughout the test via telemetry with a heart rate monitor (Polar, Kempele, Finland). A similar protocol will be used for singleleg tests, except that power will increase by 1 W every four seconds. VO2peak and will be defined as the highest oxygen consumption achieved over a 30-s period. Maximal workload (Wmax) will be the highest power output achieved during the test. The subject is deemed to have reached VO2peak if: i) the perceived exertion is >19 (Borg Scale) ii) his HR is within 5bpm of age-predicted maximal HR; iii) his RER is >1.2; and iv) a plateau has been reached in their oxygen consumption.

## DXA Scan:

Body composition (i.e. fat (%), appendicular lean mass (kg), and lean body mass (kg)) will be determined by dual-energy x-ray absorptiometry (DXA).

### **Deuterated Water:**

Deuterium is an isotope of hydrogen and is in fact already present in small amounts in the water consumed daily (i.e. 0.02%). It poses no health risk in the quantities consumed during this study, and about half of the water in the body is replaced every week. Once the participant stops drinking this water, body water will return to its normal concentration in 20-30 days. During the study, participants will be required to drink ~1 cup of deuterated water (D2O).

# Skeletal Muscle Biopsies and Analyses:

During the study, 7 muscle biopsies will be collected (days -3, 0 [4 biopsies], 1, and 2). This procedure involves the removal of a small piece of muscle tissue using a sterile hollow needle from the quadriceps muscle (*vastus lateralis*) under local aesthetic (lidocaine). A small piece of muscle (~100 mg) will be

collected at each time point. Following the biopsies, the incisions will be closed with instant medical adhesive, and wrapped with a tensor bandage. Phosphoproteomic analysis will be conducted by mass-spectrometry as previously described (41). Myofibrillar MPS will be calculated using the precursor-product equation: myofibrillar MPS =( $[E_{2b}-E_{1b}]/[E_{ic} \times f]$ ) x 100.  $E_b$ represents the enrichment of bound myofibrillar protein,  $E_{ic}$  is the average intracellular enrichment between two biopsies, and t is the tracer incorporation time in h. As we will employ 'tracer naïve' participants (had not previously participated in a study protocol where L-[ring- <sup>13</sup>C<sub>6</sub>] phenylalanine was infused), a pre-infusion blood sample will be used for the calculation of resting myofibrillar MPS (50). Myofibrillar and intracellular enrichments of L-[ring- <sup>13</sup>C<sub>6</sub>] phenylalanine will be measured as previously described (51). Integrated (i.e., days) rates of muscle protein synthesis (MPS) will be determined using the D2O method. Briefly, <sup>2</sup>H enrichment of saliva (precursor) and muscle (product) pools (relative to <sup>1</sup>H) will be determined using isotope ratio mass spectrometry and myofibrillar fractional synthetic rate determined, as previously described (52, 53).

## Diets:

Ad libitum 3-day dietary records for each participant will be collected and analyzed for baseline macronutrient intake. During the study, all food will be provided to the participants as frozen meals (Supplier: Copper County Foods), and pre-weighed and measured snack items.

## Physical activity:

Recreationally active young men (assessed through physical activity questionnaire) will be recruited. Participants will be asked to maintain their habitual activity for the duration of the study.

## Exercise Protocol:

Resistance exercise: 5 sets × 10 reps 75% 1RM leg press followed by leg extension, with 2 min recovery between sets and exercises (50).

Endurance exercise:  $4 \times 5$  min @ 65% single leg peak power with 2.5 min recovery @ 20% peak power (MacInnis 2016)

# **References**

- 1. Rennie MJ, Edwards RH, Halliday D, Matthews DE, Wolman SL, Millward DJ. Muscle protein synthesis measured by stable isotope techniques in man: the effects of feeding and fasting. Clin Sci (Lond). 1982;63(6):519-23.
- 2. Atherton PJ, Etheridge T, Watt PW, Wilkinson D, Selby A, Rankin D, et al. Muscle full effect after oral protein: time-dependent concordance and discordance between human muscle protein synthesis and mTORC1 signaling. Am J Clin Nutr. 2010;92(5):1080-8.
- 3. Morton RW, McGlory C, Phillips SM. Nutritional interventions to augment resistance training-induced skeletal muscle hypertrophy. Front Physiol. 2015;6:245.
- 4. Biolo G, Tipton KD, Klein S, Wolfe RR. An abundant supply of amino acids enhances the metabolic effect of exercise on muscle protein. Am J Physiol. 1997;273(1 Pt 1):E122-9.
- 5. Biolo G, Maggi SP, Williams BD, Tipton KD, Wolfe RR. Increased rates of muscle protein turnover and amino acid transport after resistance exercise in humans. Am J Physiol. 1995;268(3 Pt 1):E514-20.
- 6. Glynn EL, Fry CS, Drummond MJ, Dreyer HC, Dhanani S, Volpi E, et al. Muscle protein breakdown has a minor role in the protein anabolic response to essential amino acid and carbohydrate intake following resistance exercise. Am J Physiol Regul Integr Comp Physiol. 2010;299(2):R533-40.
- 7. Cermak NM, Res PT, de Groot LC, Saris WH, van Loon LJ. Protein supplementation augments the adaptive response of skeletal muscle to resistance-type exercise training: a meta-analysis. Am J Clin Nutr. 2012;96(6):1454-64.
- 8. Perry CG, Lally J, Holloway GP, Heigenhauser GJ, Bonen A, Spriet LL. Repeated transient mRNA bursts precede increases in transcriptional and mitochondrial proteins during training in human skeletal muscle. J Physiol. 2010;588(Pt 23):4795-810.
- 9. Egan B, O'Connor PL, Zierath JR, O'Gorman DJ. Time course analysis reveals gene-specific transcript and protein kinetics of adaptation to short-term aerobic exercise training in human skeletal muscle. PLoS One. 2013;8(9):e74098.
- 10. Holloszy JO. Biochemical adaptations in muscle. Effects of exercise on mitochondrial oxygen uptake and respiratory enzyme activity in skeletal muscle. J Biol Chem. 1967;242(9):2278-82.
- 11. Gibala MJ, Little JP, van Essen M, Wilkin GP, Burgomaster KA, Safdar A, et al. Short-term sprint interval versus traditional endurance training: similar initial adaptations in human skeletal muscle and exercise performance. J Physiol. 2006;575(Pt 3):901-11.
- 12. Egan B, Zierath JR. Exercise metabolism and the molecular regulation of skeletal muscle adaptation. Cell metabolism. 2013;17(2):162-84.
- 13. Nader GA, von Walden F, Liu C, Lindvall J, Gutmann L, Pistilli EE, et al. Resistance exercise training modulates acute gene expression during human skeletal muscle hypertrophy. J Appl Physiol (1985). 2014;116(6):693-702.
- 14. Mitchell CJ, Churchward-Venne TA, West DWD, Burd NA, Breen L, Baker SK, et al. Resistance exercise load does not determine training-mediated hypertrophic gains in young men. J Appl Physiol. 2012;113(1):71-7.

- 15. Campos GE, Luecke TJ, Wendeln HK, Toma K, Hagerman FC, Murray TF, et al. Muscular adaptations in response to three different resistance-training regimens: specificity of repetition maximum training zones. Eur J Appl Physiol. 2002;88(1-2):50-60.
- 16. Wilkinson SB, Phillips SM, Atherton PJ, Patel R, Yarasheski KE, Tarnopolsky MA, et al. Differential effects of resistance and endurance exercise in the fed state on signalling molecule phosphorylation and protein synthesis in human muscle. J Physiol. 2008;586(Pt 15):3701-17.
- 17. Fluck M, Hoppeler H. Molecular basis of skeletal muscle plasticity--from gene to form and function. Rev Physiol Biochem Pharmacol. 2003;146:159-216.
- 18. Vissing K, Schjerling P. Simplified data access on human skeletal muscle transcriptome responses to differentiated exercise. Sci Data. 2014;1:140041.
- 19. Mahoney DJ, Tarnopolsky MA. Understanding skeletal muscle adaptation to exercise training in humans: contributions from microarray studies. Phys Med Rehabil Clin N Am. 2005;16(4):859-73, vii.
- 20. Talanian JL, Galloway SD, Heigenhauser GJ, Bonen A, Spriet LL. Two weeks of high-intensity aerobic interval training increases the capacity for fat oxidation during exercise in women. J Appl Physiol (1985). 2007;102(4):1439-47.
- 21. Scarpulla RC. Nuclear control of respiratory chain expression by nuclear respiratory factors and PGC-1-related coactivator. Ann N Y Acad Sci. 2008;1147:321-34.
- 22. Scarpulla RC. Nuclear control of respiratory gene expression in mammalian cells. J Cell Biochem. 2006;97(4):673-83.
- 23. Scarpulla RC. Nuclear activators and coactivators in mammalian mitochondrial biogenesis. Biochim Biophys Acta. 2002;1576(1-2):1-14.
- 24. Gilde AJ, van der Lee KA, Willemsen PH, Chinetti G, van der Leij FR, van der Vusse GJ, et al. Peroxisome proliferator-activated receptor (PPAR) alpha and PPARbeta/delta, but not PPARgamma, modulate the expression of genes involved in cardiac lipid metabolism. Circ Res. 2003;92(5):518-24.
- 25. Pilegaard H, Ordway GA, Saltin B, Neufer PD. Transcriptional regulation of gene expression in human skeletal muscle during recovery from exercise. Am J Physiol Endocrinol Metab. 2000;279(4):E806-14.
- 26. Hood DA, Tryon LD, Vainshtein A, Memme J, Chen C, Pauly M, et al. Exercise and the Regulation of Mitochondrial Turnover. Prog Mol Biol Transl Sci. 2015;135:99-127.
- 27. Hood DA. Invited Review: contractile activity-induced mitochondrial biogenesis in skeletal muscle. J Appl Physiol (1985). 2001;90(3):1137-57.
- 28. Yu M, Stepto NK, Chibalin AV, Fryer LG, Carling D, Krook A, et al. Metabolic and mitogenic signal transduction in human skeletal muscle after intense cycling exercise. J Physiol. 2003;546(Pt 2):327-35.
- 29. Barres R, Yan J, Egan B, Treebak JT, Rasmussen M, Fritz T, et al. Acute exercise remodels promoter methylation in human skeletal muscle. Cell metabolism. 2012;15(3):405-11.
- 30. McGlory C, White AT, Treins C, Drust B, Close GL, Maclaren DP, et al. Application of the (gamma-32P) ATP kinase assay to study anabolic signaling in human skeletal muscle. J Appl Physiol (1985). 2014.

- 31. Drummond MJ, Fry CS, Glynn EL, Dreyer HC, Dhanani S, Timmerman KL, et al. Rapamycin administration in humans blocks the contraction-induced increase in skeletal muscle protein synthesis. J Physiol-London. 2009;587(7):1535-46.
- 32. Goodman CA, Frey JW, Mabrey DM, Jacobs BL, Lincoln HC, You JS, et al. The role of skeletal muscle mTOR in the regulation of mechanical load-induced growth. J Physiol. 2011;589(Pt 22):5485-501.
- 33. Baar K, Esser K. Phosphorylation of p70(S6k) correlates with increased skeletal muscle mass following resistance exercise. Am J Physiol. 1999;276(1 Pt 1):C120-7.
- 34. Mader S, Lee H, Pause A, Sonenberg N. The translation initiation factor eIF-4E binds to a common motif shared by the translation factor eIF-4 gamma and the translational repressors 4E-binding proteins. Mol Cell Biol. 1995;15(9):4990-7.
- 35. Raught B, Gingras AC. eIF4E activity is regulated at multiple levels. Int J Biochem Cell Biol. 1999;31(1):43-57.
- 36. Gingras AC, Gygi SP, Raught B, Polakiewicz RD, Abraham RT, Hoekstra MF, et al. Regulation of 4E-BP1 phosphorylation: a novel two-step mechanism. Genes Dev. 1999;13(11):1422-37.
- 37. Holz MK, Ballif BA, Gygi SP, Blenis J. mTOR and S6K1 mediate assembly of the translation preinitiation complex through dynamic protein interchange and ordered phosphorylation events. Cell. 2005;123(4):569-80.
- 38. Chauvin C, Koka V, Nouschi A, Mieulet V, Hoareau-Aveilla C, Dreazen A, et al. Ribosomal protein S6 kinase activity controls the ribosome biogenesis transcriptional program. Oncogene. 2014;33(4):474-83.
- 39. McGlory C, White A, Treins C, Drust B, Close GL, Maclaren DP, et al. Application of the [gamma-32P] ATP kinase assay to study anabolic signaling in human skeletal muscle. J Appl Physiol (1985). 2014;116(5):504-13.
- 40. MacInnis MJ, Haikalis ME, Martin BJ, Skelly LE, Gillen JB, Tarnopolsky MA, et al. Mitochondrial Adaptation To Training: Superior Effect Of Interval Versus Continuous Exercise When Work Is Matched: 2673 Board #196 June 3, 9: 30 AM 11: 00 AM. Med Sci Sports Exerc. 2016;48(5 Suppl 1):747.
- 41. Hoffman NJ, Parker BL, Chaudhuri R, Fisher-Wellman KH, Kleinert M, Humphrey SJ, et al. Global Phosphoproteomic Analysis of Human Skeletal Muscle Reveals a Network of Exercise-Regulated Kinases and AMPK Substrates. Cell Metab. 2015;22(5):922-35.
- 42. McCloy RA, Parker BL, Rogers S, Chaudhuri R, Gayevskiy V, Hoffman NJ, et al. Global Phosphoproteomic Mapping of Early Mitotic Exit in Human Cells Identifies Novel Substrate Dephosphorylation Motifs. Mol Cell Proteomics. 2015;14(8):2194-212.
- 43. Knowles OE, Aisbett B, Main LC, Drinkwater EJ, Orellana L, Lamon S. Resistance Training and Skeletal Muscle Protein Metabolism in Eumenorrheic Females: Implications for Researchers and Practitioners. Sports Med. 2019;49(11):1637-50.
- 44. Mitchell CJ, Churchward-Venne TA, Cameron-Smith D, Phillips SM. What is the relationship between the acute muscle protein synthesis response and changes in muscle mass? J Appl Physiol (1985). 2015;118(4):495-7.
- 45. Mitchell WK, Phillips BE, Williams JP, Rankin D, Lund JN, Wilkinson DJ, et al. The impact of delivery profile of essential amino acids upon skeletal

- muscle protein synthesis in older men: clinical efficacy of pulse vs. bolus supply. Am J Physiol Endocrinol Metab. 2015;309(5):E450-7.
- 46. Churchward-Venne TA, Burd NA, Mitchell CJ, West DW, Philp A, Marcotte GR, et al. Supplementation of a suboptimal protein dose with leucine or essential amino acids: effects on myofibrillar protein synthesis at rest and following resistance exercise in men. J Physiol. 2012;590(11):2751-65.
- 47. Burd NA, Andrews RJ, West DW, Little JP, Cochran AJ, Hector AJ, et al. Muscle time under tension during resistance exercise stimulates differential muscle protein sub-fractional synthetic responses in men. J Physiol. 2012;590(2):351-62.
- 48. Moore DR, Churchward-Venne TA, Witard O, Breen L, Burd NA, Tipton KD, et al. Protein ingestion to stimulate myofibrillar protein synthesis requires greater relative protein intakes in healthy older versus younger men. J Gerontol A Biol Sci Med Sci. 2015;70(1):57-62.
- 49. Moore DR, Tang JE, Burd NA, Rerecich T, Tarnopolsky MA, Phillips SM. Differential stimulation of myofibrillar and sarcoplasmic protein synthesis with protein ingestion at rest and after resistance exercise. J Physiol. 2009;587(Pt 4):897-904.
- 50. McGlory C, Wardle SL, Macnaughton LS, Witard OC, Scott F, Dick J, et al. Fish oil supplementation suppresses resistance exercise and feeding-induced increases in anabolic signaling without affecting myofibrillar protein synthesis in young men. Physiol Rep. 2016;4(6).
- 51. Churchward-Venne TA, Burd NA, Mitchell CJ, West DW, Philp A, Marcotte GR, et al. Supplementation of a suboptimal protein dose with leucine or essential amino acids: effects on myofibrillar protein synthesis at rest and following resistance exercise in men. J Physiol. 2012;590(Pt 11):2751-65.
- 52. McGlory C, Gorissen SHM, Kamal M, Bahniwal R, Hector AJ, Baker SK, et al. Omega-3 fatty acid supplementation attenuates skeletal muscle disuse atrophy during two weeks of unilateral leg immobilization in healthy young women. FASEB J. 2019;33(3):4586-97.
- 53. Wilkinson DJ, Franchi MV, Brook MS, Narici MV, Williams JP, Mitchell WK, et al. A validation of the application of D(2)O stable isotope tracer techniques for monitoring day-to-day changes in muscle protein subfraction synthesis in humans. Am J Physiol Endocrinol Metab. 2014;306(5):E571-9.